CLINICAL TRIAL: NCT04457323
Title: Comparison of Efficacy and Safety of S-Metoprolol XR 25-50 mg Tablets and Metoprolol Zok 50-100 mg Tablets in Hypertensive Patients.
Brief Title: S-Metoprolol XR 25-50 mg Tablets vs Metoprolol Zok 50-100 mg Tablets in Hypertension Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Neutec Ar-Ge San ve Tic A.Ş (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEU-03.17
Record Dates: First submitted 2020-06-25; First posted 2020-07-07 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Metoprolol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental): S-Metoprolol XR 25 mg Film Coated Tablets (first four weeks) S-Metoprolol XR 50 mg Film Coated Tablets (second four weeks)
  Interventions: Drug: Metoprolol
- REFERENCE (Active Comparator): Beloc® (Metoprolol) Zok 50 mg Controlled Release Film Tablets (first four weeks) Beloc® (Metoprolol) Zok 100 mg Controlled Release Film Tablets (second four weeks)
  Interventions: Drug: Metoprolol

INTERVENTIONS:
Drug: Metoprolol — S-Metoprolol XR 25 mg and 50 mg Film Coated Tablets
  Other Names: S-metoprolol
  Arms: Test
Drug: Metoprolol — Beloc® (Metoprolol) Zok 50 mg and 100 mg Controlled Release Film Tablets
  Arms: REFERENCE

SUMMARY:
The aim of this study is to compare the efficacy and safety of S-Metoprolol XR 25 and 50 mg Film Coated Tablets and Beloc® (Metoprolol) Zok 50 and 100 mg Controlled Release Film Tablets administered once daily, in the treatment of hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients: between the ages of 18-70,
* Stage 1 and 2 hypertension patients who have not received any antihypertensive treatment in the past month * (≥ 140 mmHg SKB <180 mmHg, ≥ 90 mmHg DKB <110 mmHg,
* Patients with minute heart rate ≥ 70 / min,
* Patients followed up with outpatient treatment,
* Patients who give written informed consent without any influence, (Stage 1 Hypertension; SKB: 140-159 mmHg and DKB: 90-99 mmHg, Stage 2 Hypertension; SKB: 160--179 mmHg and DKB: 100--109 mmHg)

Exclusion Criteria:

* Pregnant patients or breastfeeding mothers or women with childbearing potential who do not use any effective contraceptive methods,
* Patients with allergies or hypersensitivity to betabloker drugs,
* Patients who have received antihypertensive treatment in the past month,
* Patients with secondary hypertension,
* Patients who were followed up for the following diseases from the beginning of the study until the last 12 months,

  * Severe hypertension (SKB> 180 mmHg and / or DKB> 110 mmHg),
  * Myocardial infarction,
  * NYHA stage 2-4 heart failure,
  * Patients with a history of cerebrovascular disease, previous ischemic attack, encephalopathy,
  * Patients undergoing percutaneous coronary intervention or coronary artery bypass surgery,
  * 2nd or 3rd degree heart block or symptomatic arrhythmia without pacemaker,
  * Clinically significant heart valve disease,
  * Simultaneous life-threatening potential or symptomatic arrhythmia,
  * Simultaneous unstable angina pectoris,
  * Type 1 DM,
  * Atrial fibrillation,
  * Uncontrollable Type 2 DM (HbA1C> 7%),
* Patients with significant liver disease (initial ALT, AST> 2xULN, esophageal varices, portocaval shunt),
* Patients with significant kidney disease (GFR <60 ml / min according to the Cockcroft-Gault formula),
* Patients with volume depletion,
* Patients with pancreatic disease,
* Patients with gastrointestinal disease affecting absorption,
* Drug/substance and alcohol abuse in the last 12 months,
* Patients with central nervous system disease and using drugs for this reason,
* A history of incompatibility with medical regimens, or patients' unwillingness to comply with the study protocol,
* Patients directly involved in the management of this protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2022-01-15 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure between 0-4 weeks of treatment | 4-weeks

SECONDARY OUTCOMES:
Change in systolic blood pressure between 0-8 weeks of treatment. | 8-weeks
Change in diastolic blood pressure between 0-8 weeks of treatment. | 8-weeks
Change in diastolic blood pressure between 4-8 weeks of treatment. | 4-weeks
Change in sistolic blood pressure between 4-8 weeks of treatment. | 8-weeks
Treatment response rates | 4-weeks
  Target blood pressure values were determined by decreasing more than 20mmHg in systolic blood pressure and / or decreasing more than 10mmHg in diastolic pressure (under systolic 140 mmHg, below diastolic 90 mmHg).

IPD SHARING:
Plan to Share IPD: Undecided